CLINICAL TRIAL: NCT05390944
Title: An Open-label, Randomized, Single-dose, Two-way Crossover Bioequivalence Study to Compare Two Strengths (10 mg and 20 mg) of IMP4297 Capsules in Healthy Chinese Subjects Under Fasting Condition
Brief Title: An BE Study to Compare 10mg & 20mg of IMP4297 Capsules in Healthy Chinese Subjects Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Impact Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IMP4297-110-1
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor
MeSH Terms: interventions — senaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IMP4297 first 5*20mg then 10*10mg (Experimental): Single oral dose of IMP4297 administered under fasting conditions 5*20 mg capsules in first intervention period and 10*10 mg capsules in second intervention period (after washout period: at least 7 days)
  Interventions: Drug: IMP4297(20mg); Drug: IMP4297(10mg)
- IMP4297 first 10*10mg then 5*20mg (Experimental): Single oral dose of IMP4297 administered under fasting conditions 10*10 mg capsules in first intervention period and 5*20 mg capsules in second intervention period (after washout period: at least 7 days)
  Interventions: Drug: IMP4297(20mg); Drug: IMP4297(10mg)

INTERVENTIONS:
Drug: IMP4297(20mg) — Single oral dose of IMP4297 administered under fasting conditions 5*20 mg capsules in first intervention period and 10*10 mg capsules in second intervention period (after washout period: at least 7 days)
Drug: IMP4297(10mg) — Single oral dose of IMP4297 administered under fasting conditions 10*10 mg capsules in first intervention period and 5*20 mg capsules in second intervention period (after washout period: at least 7 days)

SUMMARY:
An open-label, randomized, single-dose, two-way crossover bioequivalence study to compare two strengths (10 mg and 20 mg) of IMP4297 capsules in healthy Chinese subjects under fasting condition.

DETAILED DESCRIPTION:
An open-label, randomized, single-dose, two-way crossover bioequivalence study is designed to determine whether IMP4297 capsules 100 mg (5 × 20 mg strength) and IMP4297 capsules 100 mg (10 × 10 mg strength) are bioequivalent in healthy Chinese male subjects under fasting condition.

28 subjects (at least 22 completed) are planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for the study

1. The subject fully understands the objective, nature, method of the trial and possible adverse reactions, voluntarily acts as a subject, signs the informed consent form before any study procedure, and ensures that any procedure is performed by himself/herself.
2. Healthy Chinese male subjects aged 18 to 55 years (inclusive) at Screening.
3. Body mass index (BMI) between 19.0 and 26.0 kg/m2 (inclusive); body weight ≥50.0 kg.
4. Subject is able to communicate well with the Investigator and understands and adheres to the requirements of the study.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria is not allowed to participate in the study:

1. Subjects with diseases with abnormal clinical manifestations requiring exclusion, including but not limited to diseases of nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolism and bone system.
2. History of allergic diseases (including drug allergies and food allergies, etc.), and allergy to IMP4297 capsules or any component of the product.
3. History of dysphagia or any gastrointestinal disease affecting drug absorption (as judged by the investigator).
4. Subjects having experienced surgery within 3 months prior to screening, or having a surgery planned during the study period, and having received any surgery that may affect drug absorption (e.g., gastrectomy).
5. Subjects who cannot tolerate venipuncture and who ever fainted during injection or at sight of blood.
6. Lactose intolerance (those who had diarrhea after drinking milk).
7. History of drug abuse within 6 months prior to screening, or a positive result on the urine drug screen (screening or baseline).
8. Subjects who drink more than 14 units of alcohol (1 unit of alcohol = 360 mL of beer, 150 mL of wine, or 45 mL of liquor) per week within 3 months prior to screening, or have a positive breath alcohol test (screening or baseline), or cannot abstain from alcohol during the trial.
9. Subjects who smoke more than 5 cigarettes per day on average within 3 months prior to screening, or cannot stop using any tobacco products during the trial.
10. Subjects who consumed excessive amount of tea, coffee, and/or caffeine-rich beverages (more than 8 cups, 1 cup = 250 mL) per day on average during the 3 months prior to screening.
11. Subjects who have participated in the clinical trial of other study drug/device within 3 months before the first administration of the study drug, or have participated in 3 or more clinical trials of drugs/devices in the past year; if the half-life of other study drugs is longer, the longer time interval is required, that is, 5 half-lives of the drug.
12. Blood donation with blood components or significant blood loss (≥ 200 mL) within 3 months prior to screening; blood transfusion or use of blood products and blood biological products within 3 months prior to screening.
13. Subjects who have received live vaccination within 4 weeks prior to screening.
14. Used any drugs [e.g. barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; SSRI antidepressants, cimetidine, macrolides, nitroimidazoles, sedative hypnotics, fluoroquinolones, antihistamines, antiviral drugs (such as saquinavir, etc.), calcium antagonists (such as diltiazem, verapamil, etc.), rifamycins (such as rifampicin, etc.)] that inhibit or induce hepatic metabolism of drugs within 28 days prior to taking study drug. If the half-life of a prior medication is longer, the required time interval will also be prolonged, that is, 5 half-lives of the drug, e.g. a 5-week washout period for phenobarbital.
15. Used prescription drugs, over-the-counter drugs, dietary supplements, or Chinese herbal medicines within 14 days prior to the first dose of study drug. If the half-life of a prior medication is longer, the required time interval will also be prolonged, that is, 5 half-lives of the drug. For over-the-counter medications that are not considered to affect the overall outcome of the study, limited use is permitted on a case-by-case basis after approval by the Sponsor and the Investigator.
16. Positive for any of the hepatitis B surface antigen, hepatitis B core antibody, hepatitis C virus antibody, anti-human immunodeficiency virus antibody, or treponema pallidum antibody tests.
17. Subjects with clinically significant abnormalities in vital signs (blood pressure, pulse and body temperature), complete physical examination, laboratory tests (hematology, blood chemistry and urinalysis) at screening as judged by the investigator; refer to normal range (including critical values) for vital signs: sitting systolic pressure 90-140 mmHg, diastolic pressure 60-90 mHg, pulse 60-100 beats/min, body temperature (ear temperature) 35.7-37.9°C, subjected to the comprehensive judgment by the investigator.
18. Corrected QT interval (corrected according to Fridericia's formula, QTcF = QT/RR1/3) from 12-lead ECG in supine position in the resting state (at least 5 min) at screening > 450 msec or QRS complex > 120 msec. If QTcF exceeds 450 msec or QRS exceeds 120 msec, 2 additional ECGs should be repeated, and the average of the 3 measured QTcF or QRS values are judged by the investigator to be clinically significant abnormalities.
19. Subjects who cannot stop strenuous exercise within 48 hours before the first dose of the study drug and during the trial.
20. Consumed any alcoholic, caffeine, chocolate, xanthine-rich food or beverage within 48 h before the first administration of the study drug; or unable to fast from these products during the trial.
21. Subjects who cannot fast from grapefruit or grapefruit-related citrus (e.g., pomelo) fruits or juices within 7 days prior to the first dose of study drug and during the trial.
22. Subjects or their partners have fertility plan during the whole process of the study and within 90 days after the last dose of the study drug, or are unwilling to take effective contraceptive measures (Appendix 1), or have sperm donation plan.
23. Unwilling or unable to follow the protocol-specified lifestyle guidelines (e.g., dietary restrictions and activity requirements).
24. Other acute or chronic medical or psychiatric condition that, in the judgment of the investigator, would make the subject inappropriate for this study, might increase the risk associated with participation in this study, or might interfere with the interpretation of study results.
25. Other subjects who are not suitable to participate in the clinical trial as judged by the investigator.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Cmax | 0-72 hours
  Maximum concentration. In each cycle, blood PK samples are collected at 0 hour (within 1 hour pre-dose) and 0.25 hour, 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 4 hour, 5 hour, 6 hour, 8 hour, 10 hour, 12 hour, 24 hour, 48 hour and 72 hour post-dose for analysis of plasma IMP4297 concentrations, with quiet rest for 5 minutes after blood collection.
AUC0-last | 0-72 hours
  area under the drug concentration-time curve from time 0 to the last time with quantifiable concentration. In each cycle, blood PK samples are collected at 0 hour (within 1 h pre-dose) and 0.25 hour, 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 4 hour, 5 hour, 6 hour, 8 hour, 10 hour, 12 hour, 24 hour, 48 hour and 72 hour post-dose for analysis of plasma IMP4297 concentrations, with quiet rest for 5 minutes after blood collection.
AUC0-inf | 0-72 hours
  area under the curve from time 0 to infinity. In each cycle, blood PK samples are collected at 0 hour (within 1 hour pre-dose) and 0.25 hour, 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 4 hour, 5 hour, 6 hour, 8 hour, 10 hour, 12 hour, 24 hour, 48 hour and 72 hour post-dose for analysis of plasma IMP4297 concentrations, with quiet rest for 5 minutes after blood collection.

CONTACTS AND LOCATIONS:
Overall Officials: Chuanling Li, Principal Investigator — Xuzhou Central Hospital
Locations (1):
- Xuzhou Central Hospital, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No